CLINICAL TRIAL: NCT02239900
Title: Phase I/II Trial of Ipilimumab (Immunotherapy) and Hypofractionated Stereotactic Radiation Therapy in Patients With Advanced Solid Malignancies
Brief Title: Ipilimumab and Stereotactic Body Radiation Therapy (SBRT) in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0882; NCI-2015-00042 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Liver Cancer; Lung Cancer
Keywords: Liver Cancer; Lung Cancer; Adrenal Gland; Metastasis; Advanced Solid Malignancies; Ipilimumab; Yervoy; BMS-734016; MDX010; Stereotactic Body Radiation Therapy; SBRT; XRT
MeSH Terms: conditions — Liver Neoplasms; Lung Neoplasms; Neoplasm Metastasis | interventions — Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 Liver: Concurrent (early) Ipilimumab and SBRT (Experimental): Participants with at least 1 liver metastasis - Treatment Group 1: Ipilimumab 3 mg/kg by vein on Day 1 of all 21 day cycles for a total of 4 doses. SBRT 50 Gy in 4 fractions to 1 - 4 liver lesion(s) on Days 1 - 4 of Cycle 1.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Group 2 Liver: Sequential (late) Ipilimumab and SBRT (Experimental): Participants with at least 1 liver metastasis - Treatment Group 2: Ipilimumab 3 mg/kg by vein on Day 1 of Cycles 1 and 2. After SBRT treatment, Ipilimumab given on Day 1 of Cycles 3 and 4. Each cycle is 21 days. SBRT 50 Gy in 4 fractions to 1 - 4 liver lesion(s) on Days 29 - 33 of each 21 day cycle.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Group 3 Lung: Concurrent (early) Ipilimumab and SBRT (Experimental): Participants with at least 1 lung metastasis - Treatment Group 3: Ipilimumab 3 mg/kg by vein on Day 1 of all 21 day cycles for a total of 4 doses. SBRT 50 Gy in 4 fractions to 1 - 4 lung lesion(s) on Days 1 - 4 of Cycle 1.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Group 4 Lung: Sequential (late) Ipilimumab and SBRT (Experimental): Participants with at least 1 lung metastasis - Treatment Group 4: Ipilimumab 3 mg/kg by vein on Day 1 of Cycles 1 and 2. After SBRT treatment, Ipilimumab given on Day 1 of Cycles 3 and 4. Each cycle is 21 days. SBRT 50 Gy in 4 fractions to 1 - 4 lung lesion(s) on Days 29 - 33 of each 21 day cycle.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Group 5 Liver/Lung Metastasis: (late) Ipilimumab and SBRT (Experimental): Participants with 1 liver or lung metastasis - Treatment Group 5: Ipilimumab 3 mg/kg by vein on Day 1 of Cycle 1. After SBRT treatment, Ipilimumab given on Day 1 of Cycles 2 - 4. Each cycle is 21 days. SBRT 60 Gy in 10 fractions to 1 - 4 lung, liver, or adrenal lesion (s) on Days 1 - 5 and Days 9 - 12 of Cycle 1.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Thyroid Expansion Cohort (Experimental): Participants enrolled in this arm treated to a total dose of 50 Gy in 4 fractions, 60 Gy in 10 fractions, or 20 Gy in 5 fractions with stereotactic radiotherapy to a liver or lung lesion. The choice of radiation dose will be at the discretion of the treating radiation oncologist.
  Participants receive Ipilimumab every 21 days for a total of 4 doses.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Ipilimumab — Treatment Group 1 and 3: Ipilimumab 3 mg/kg by vein on Day 1 of all 21 day cycles for a total of 4 doses.
  Treatment Group 2 and 4: Ipilimumab 3 mg/kg by vein on Day 1 of Cycles 1 and 2. After SBRT treatment, Ipilimumab given on Day 1 of Cycles 3 and 4.
  Treatment Group 5: Ipilimumab 3 mg/kg by vein on Day 1 of Cycle 1. After SBRT treatment, Ipilimumab given on Day 1 of Cycles 2-4
  Other Names: Yervoy; BMS-734016; MDX010
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Treatment Group 1 and 3: SBRT 50 Gy in 4 fractions to 1 - 4 liver lesion(s) on Days 1 - 4 of Cycle 1.
  Treatment Group 2 and 4: SBRT 50 Gy in 4 fractions to 1-4 liver lesion(s) on Days 29 - 33 of each 21 day cycle.
  Treatment Group 5: SBRT 60 Gy in 10 fractions to 1 - 4 lung, liver, or adrenal lesion (s) on Days 1 - 5 and Days 9 - 12 of Cycle 1.
  Other Names: SBRT; XRT

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of ipilimumab and stereotactic body radiation therapy (SBRT). The safety and effectiveness of these treatments given consecutively will also be studied.

This is an investigational study. SBRT is FDA approved for the control of metastatic and primary tumors. Ipilimumab is FDA approved and commercially available for the treatment of metastatic melanoma that cannot be removed with surgery. The use of SBRT with ipilimumab is investigational. The study doctor can explain how the study drug is designed to work.

Up to 120 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

Participants on this study are enrolled into Phase 1 (Dose De-Escalation, or Dose-Finding) or Phase 2 (Dose Expansion), based on when they join the study.

Phase 1: Dose De-Escalation:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 5 groups based on the type of disease you have.

* If you are in Groups 1 or 3, you will receive SBRT and 1 dose of ipilimumab within a few days after your SBRT treatment, and then you will receive 3 more doses of ipilimumab.
* If you are in Groups 2, 4, or 5, you will receive 2 doses of ipilimumab, SBRT, and then 2 more doses of ipilimumab.

If you are in Group 5, SBRT will be given over a longer period of time (more days or weeks).

All participants will receive the same dose level of ipilimumab.

You will be given a separate consent form explaining SBRT and its risks.

In each group, 3 participants will be enrolled at the first dose level. If no more than 1 participant has intolerable side effects, up to 3 more participants will be enrolled at that dose level. If no intolerable side effects are seen at that dose level, that is considered the highest tolerated dose.

If enough intolerable side effects are seen at the assigned dose level, the total dose amount of radiation given in any group may be lowered up to 2 times.

Phase 2: Dose Expansion:

Once the highest tolerated dose combination is found in each study group, up to 14 more participants will be enrolled at that dose level combination in each group.

Study Drug Administration:

Each study cycle is 21 days.

If you are in Groups 1 or 3 (early ipilimumab and SBRT), you will receive ipilimumab by vein over about 90 minutes on Day 1 of all cycles. You will also receive SBRT over about 30-45 minutes on Days 1-4 of Cycle 1.

If you are in Groups 2 or 4 (late ipilimumab and SBRT), you will receive ipilimumab by vein over about 90 minutes on Day 1 of Cycles 1 and 2 and then SBRT on Days 29-33. After your SBRT treatment, you will take ipilimumab on Day 1 of Cycles 3 and 4.

If you are in Group 5 (late ipilimumab and SBRT), you will receive ipilimumab on Day 1 of Cycle 1 and SBRT over about 30-45 minutes on Days 1-5 and Days 9-12 of Cycle 1. After your SBRT treatment, you will take ipilimumab on Day 1 of Cycles 2-4.

You will be given standard drugs to help decrease the risk of side effects and to help support your immune system. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

During Week 1 of all cycles and Week 2 of Cycle 2:

* You will have a physical exam, including measurement of your weight.
* Blood (about 1 tablespoon) will be drawn for routine tests.

During Week 3 of Cycles 2 and 4, you will have an MRI, CT scan, and/or PET/CT scan to check the status of the disease.

If you are in Phase 2, during Week 3 of each cycle, blood (about 2 teaspoons) may be drawn for biomarker testing, if the doctor thinks it is safe.

You may have a chest scan if the doctor thinks it is needed.

Length of Study:

You may receive up to 4 cycles of treatment with ipilimumab and SBRT. About 8 weeks after you have completed Cycle 4, if the size of the tumor does not change or it gets smaller while you are receiving therapy, you may be able to continue to receive ipilimumab and/or radiation. The study doctor will discuss this option with you.

You will no longer be able to receive treatment if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after you have completed the follow-up visits.

Follow-Up:

About 30 days after your last dose of ipilimumab and then every 3 months after that for up to 2 years, you will come to the clinic for follow-up visits. At these visits:

* You will have a physical exam, including measurement of your weight..
* Blood (about 1 tablespoon) be drawn for routine tests.
* Blood (about 2 teaspoons) may be drawn for biomarker testing, if the doctor thinks it is safe.
* Urine will be collected for routine tests.
* You will have an MRI, CT scan, and/or PET/CT scan to check the status of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histological confirmation of metastatic cancer with at least one metastatic or primary lesion in the liver, lung, or adrenal gland.
2. Patients who have completed previous systemic therapies 5 drug half-lives or 4-weeks prior to enrollment on study, whichever is shorter. Note: patients with anaplastic thyroid will be waived from this inclusion criteria given the rapid trajectory of their disease.
3. All patients must have at least one metastatic or primary lesion within the lung or liver located in an anatomical location amenable to SBRT treatment with 50 Gy in 4 fractions, or if not, with either a lung, liver, or adrenal lesion treatable to 60 Gy in 10 fractions.
4. Repeat radiation in fields previously radiated will be allowed at the discretion of the treating physician.
5. Age >/= 18 years
6. ECOG performance status </=2 (Karnofsky >60%).
7. Patients must have normal organ and marrow function as defined below: * Total bilirubin </= 2.0 mg/dL. (Does NOT apply to patients with Gilbert's Syndrome) * Aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT)/ Alanine Aminotransferase (ALT) Serum Glutamic-Pyruvic Transaminase (SGPT) <2.5 X institutional upper limit of normal (patients with liver involvement will be allowed </= 5.0 X institutional upper normal limit) *WBC >/= 2500/uL, ANC >/= 1000/uL *Platelets >/= 75K *Hemoglobin >/= 9g/dL *Creatinine </= 2.0 x ULN
8. Patients must be willing and able to review, understand, and provide written consent before starting therapy.
9. Patients with brain metastasis will be included as long as they are free of neurologic symptoms related to metastatic brain lesions and who do not require or receive systemic corticosteroid therapy in the 14 days prior to beginning ipilimumab therapy
10. Patients that have previously progressed on immunotherapy such as ipilimumab will be eligible.

Exclusion Criteria:

1. Serious autoimmune disease at the discretion of the treating attending: Patients with a history of active serious inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.
2. Active diverticulitis, intra-abdominal abscess, Gastrointestinal (GI) obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
3. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of Adverse Events: (AE's) e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Known active HIV, Hepatitis B, or Hepatitis C that has not been documented to be cured.
6. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab).
7. Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids while receiving ipilimumab (as long as steroid replacement is significantly greater than what is required for physiologic replacement, i.e. in hypothyroidism).
8. Pregnant women are excluded from this study. Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation. Acceptable forms of birth control include: Birth control pills plus a barrier method, such as a condom or diaphragm, Intrauterine devices (IUD) plus a barrier method, Implantable or injectable birth control (such as NorplantR or epo-ProveraR) started at least 3 months before joining the study, plus a barrier method, or Double-barrier method, such as a condom when used in combination with a diaphragm. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician.
9. History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician.
10. Prior allogeneic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ipilimumab and Stereotactic Body Radiation Therapy (SBRT) | Third week of second, 21 day cycle
  MTD defined as highest dose level with less than 2 patients with dose limiting toxicity (DLT) out of at least six patients in the cohort. All enrolled participants will be considered in the DLT analysis. If at any time more than or equal to one third (33%) of participants at a dose level experience DLT, the MTD will be reassessed and the next lowest dose level for the combination therapy considered the MTD.

SECONDARY OUTCOMES:
Response Rate of Ipilimumab and Stereotactic Body Radiation Therapy (SBRT) | 30 days after last dose of Ipilimumab
  Response and progression evaluated using guidelines proposed by the Immune Related Response Criteria (irRC). Patients with measurable disease also assessed using standard Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and World Health Organization (WHO) treatment response criteria. Complete Response (irCR): complete disappearance of all lesions (whether measurable or not, and no new lesions) confirmation by a repeat, consecutive imaging assessment no less than 4 wk from the date first documented. Partial Response (irPR): decrease in tumor burden ≥50% relative to baseline confirmed by a consecutive imaging assessment at least 4 wk after first documentation. Progressive Disease (irPD): increase in tumor burden ≥25% relative to nadir (minimum recorded tumor burden) confirmation by a repeat, consecutive imaging assessment no less than 4 wk from date first documented.

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] He K, Hong DS, Tang C, Sezen D, Cox L, Maleki A, Bertolet G, Nguyen QN, Comeaux NI, Schuda L, Chen D, Welsh JW. Five-year overall survival with ipilimumab and stereotactic ablative radiotherapy for metastatic disease. Radiother Oncol. 2023 Jun;183:109618. doi: 10.1016/j.radonc.2023.109618. Epub 2023 Mar 13. PMID 36921766
- [Derived] Chen D, Menon H, Verma V, Guo C, Ramapriyan R, Barsoumian H, Younes A, Hu Y, Wasley M, Cortez MA, Welsh J. Response and outcomes after anti-CTLA4 versus anti-PD1 combined with stereotactic body radiation therapy for metastatic non-small cell lung cancer: retrospective analysis of two single-institution prospective trials. J Immunother Cancer. 2020 Jan;8(1):e000492. doi: 10.1136/jitc-2019-000492. PMID 31996395
- [Derived] Cabanillas ME, McFadden DG, Durante C. Thyroid cancer. Lancet. 2016 Dec 3;388(10061):2783-2795. doi: 10.1016/S0140-6736(16)30172-6. Epub 2016 May 27. PMID 27240885
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org